Implementation Intervention to Improve Care for Unhealthy Alcohol Use (CDA 20-057)

NCT04565899

January 6, 2021

#### VA VERBAL CONSENT

# Veteran Perspectives on Alcohol-Related Care in VA Primary Care

[PRIOR TO COMMENCING INTERVIEW, INTERVIEWER READS]

Thank you for considering participating in this study. The purpose of this study is to learn about Veterans' experiences with receiving alcohol-related care at VA \*\*\*\* primary care offices. Through this study, we hope to improve the quality of care being delivered to Veterans with unhealthy alcohol use. You have been selected to participate in this study because you have received primary care services at VA \*\*\*\* campus and have drank alcohol in the past year. You should have received some mail from this study, which included an Information Statement that described what was involved, including risks and benefits.

Did you have a chance to review the Information Statement?

**If YES:** Before we begin the formal consent process, do you have any questions about the study or the procedures?

**If NO:** OK, as part of the consent process I will review what was included in the Information Statement. You can stop me at any time to ask questions. If you have additional questions after this interview, you can contact anyone on the Information Statement with the contact number provided. Do you have any questions at this time?

**STUDY DESCRIPTION:** Your participation in this study involves a 30-minute-1 hour interview and a short demographic questionnaire. Participation is completely voluntary and your answers will be held confidential. In this interview, we will ask you to recall your experiences receiving alcohol-related care at VA \*\*\*\* primary care offices. There are no right or wrong answers to any of our questions. You may skip any question that you do not feel comfortable answering or stop the interview at any time. You will be paid \$35 for your time.

You may not directly benefit from participating in this study. However, by participating, you will be making a meaningful contribution in helping us learn about improving care for Veterans with unhealthy alcohol use

In order to make sure we capture all of your responses, we will be audio-recording this interview. We also need to record you providing consent to participate in this study. After the interview, the audio-recorder

Version 2; 01/06/2021 1 of 3

### **Veteran Perspectives on Alcohol-Related Care**

#### RESEARCH VERBAL CONSENT

will be stored in a locked cabinet when not in use and will be accessible only to authorized study staff. If we are recording the interview with a remote secure VA-approved conferencing system, such as Microsoft Teams, the recording will be stored on the secure VA network with restricted access. Your audio-recording and transcript will be retained in accordance with the Veterans Health Administration (VHA) Records Control Schedule, or longer, if required by other Federal regulations.

Your privacy is important to us. Although there are many procedures in place to protect your privacy, there is the potential risk that your information could be released by mistake. We will not place personal identifiers (such as your name, address, and social security number) on any study data, including the transcript. Instead, we will assign a study code whenever possible to identify your information. Study data and transcripts will be stored on the secure VA network with restricted access.

Once this study is completed, we will not use the study code linking you to your data for any additional research. We will store the code linking you to your data separate from the study data in a secure database or in a locked filing cabinet in accordance with the VHA Records Control Schedule. If you have any questions or concerns about the research, your rights, or a possible research-related adverse event, you may contact the study team at: \*\*\*\*.

Do you have any questions regarding the study?

Okay, if we have answered all your questions, do you consent to participating in this research study?

If NO: Thank you for your time.

**If YES:** Thank you for consenting to participate.

If YES: Proceed to the Interview Guide (consent for audio-recording and begin interview).

Version 2; 01/06/2021 2 of 3

## RESEARCH VERBAL CONSENT

| TO BE COMPLETED BY THE INTERVIEWER | |
|------------------------------------------------------|-------------|
| STUDY ID: | |
| Participant consents to participate in study: Yes No | |
| Signature of Person Obtaining Consent | <b>Date</b> |
| Print Name of Person Obtaining Consent | |

Version 2; 01/06/2021 3 of 3